CLINICAL TRIAL: NCT05313685
Title: A Feasibility Double-Blinded, Randomized Study of Educational Materials for Hiccups
Brief Title: Educational Materials for Hiccups
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Aminah Jatoi, M.D., Principal Investigator, Mayo Clinic
Other Study IDs: 21-012057
Record Dates: First submitted 2022-03-28; First posted 2022-04-06 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Hiccup
MeSH Terms: conditions — Hiccup

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mayo Clinic hiccup educational materials
- Mayo Clinic hiccup educational materials + updated supplementary content

SUMMARY:
This is a research study about hiccup educational materials. The purpose of this study is to learn whether this type of research can be done.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age.
* Hiccups in the 4 weeks prior to phone contact (patient must confirm).
* Able to speak and read English.
* Has an e-mail address.

Exclusion Criteria:

- Individuals < 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have had hiccups in the preceding four weeks or patients who might be at risk for hiccups based on drug exposure (for example, recent dexamethasone exposure).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
Feasibility of enrollment | 5 months
  This is a feasibility study that seeks to enroll 20 patients with hiccups in 5 months from the start of trial recruitment.

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials